CLINICAL TRIAL: NCT03919253
Title: Pyrotinib in Combination With Nab-paclitaxel in Patients With HER2-positive Advanced Breast Cancer: an Exploratory Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBBL-01
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pyrotinib maleate tablets+nab-paclitaxel (Experimental): pyrotinib maleate tablets: 400mg orally once daily continunously; nab-paclitaxel: 125mg/m2 iv d1、8 of each 21 day cycle, 6cycles.
  Interventions: Combination Product: pyrotinib maleate tablets+nab-paclitaxel

INTERVENTIONS:
Combination Product: pyrotinib maleate tablets+nab-paclitaxel — pyrotinib maleate tablets: 400mg orally once daily continunously nab-paclitaxel: 125mg/m2 iv d1、8 of each 21 day cycle, 6cycles.

SUMMARY:
This clinical trial aim to evaluate the efficacy and safety of Pyrotinib in combination with nab-paclitaxel in patients with HER2-positive advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18-70 years old，female; 2. Pathologically confirmed HER2-positive invasive breast cancer by local laboratory with the following requirements: HER2 overexpressed or amplified (immunohistochemistry of 3+ or HER2 gene amplification by in situ hybridization) 3. Imaging examination confirmed recurrent/metastatic breast cancer； 4. Patients must have previous treatment with trastuzumab more than 9 weeks; 5. Untreated for metastatic/metastatic disease (except for endocrinotherapy); 6. Patients with at least one measurable lesions by RECIST version 1.1； 7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2； 8. Life expectancy greater than or equal to 3 months; 9. Participants must have normal organ and marrow function as described below： Absolute neutrophil count≥1.5×109/L; Platelets≥90×109/L; Hemoglobin ≥90g/L； Total bilirubin ≤ 1.5 X institutional upper limit of normal (ULN)； ALT and AST≤2*ULN, but ≤5*ULN with liver metastases; BUN and Cr≤1.5×ULN or creatinine clearance ≥50ml/min Left ventricular ejection fraction (LVEF) ≥ 50% 10. Doctors believe that treatment can bring benefits to patients； 11. Participants were willing to join in this study, and written informed consent.

Exclusion Criteria:

* 1. A variety of factors influencing oral drugs (after resection of the gastrointestinal, unable to swallow, Chronic diarrhea, intestinal obstruction); 2. Patients with other malignant tumors within 5 years (except for skin basal cell carcinoma and cervical carcinoma in situ); 3. History of psychiatric drugs abuse or patients with mental disorders; 4. Pregnant or lactating women; 5. Less than 4 weeks from the last clinical trial 6. The researchers think inappropriate.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-04-30 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival(PFS) | three years
  Baseline to measured date of progress or death from any cause

SECONDARY OUTCOMES:
Objective response rate (ORR) | three years
  Baseline to measured stable disease
Clinical Benefit Rate (CBR) | three years
  The percentage of subjects with Complete Response, Partial Response, or Stable Disease at least 24 weeks
Disease control rate(DCR) | three years
  Rate of the patients with disease control
Overall survival (OS) | up to death
  Baseline to measured date of death from any cause
Safety (number of Participants with adverse events) | three years
  Adverse events Toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. The number of Participants with adverse events will be recorded at each treatment visit.